CLINICAL TRIAL: NCT04705844
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of Adalimumab (Humira) or Placebo in Patients With Mild-Moderate COVID-19
Brief Title: Study of Adalimumab or Placebo in Patients With Mild to Moderate COVID-19 (COMBAAT)
Acronym: COMBAAT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: study withdrawn prior to screening subjects
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: Pharm-Olam, LLC (Industry); Chemical, Biological, Radiological, and Nuclear Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A21-070
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Mild to Moderate COVID-19
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive a single dose of adalimumab or placebo. Subjects will receive standard care of therapy (per study site written policies or guidelines) together with adalimumab or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adalimumab (Experimental): single dose of adalimumab(160 mg administered as 4×40 mg subcutaneous [SC] injections at separate sites on the thigh or abdomen
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): single dose of placebo (administered as 4×40 mg subcutaneous [SC] injections at separate sites on the thigh or abdomen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — adalimumab (160 mg administered as 4×40 mg subcutaneous [SC] injections at separate sites on the thigh or abdomen)
  Other Names: Humira
  Arms: Adalimumab
Drug: Placebo — placebo (4 SC injections of equal volume administered at separate sites on the thigh or abdomen)
  Arms: Placebo

SUMMARY:
Clinical study of Humira (adalimumab) or placebo in subjects with mild-moderate COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Subject (or their legally authorized representative) is willing and able to provide written informed consent prior to performing study procedures.
* Understands and agrees to comply with planned study procedures.
* Male or non-pregnant female adult ≥60 and ≤ 80years of age OR male or non-pregnant female adult ≥40 and ≤80 years, with one or more of the following risk factors (asthma, diabetes, hypertension, obesity [body mass index >30], cardiovascular disease).
* Has a laboratory-confirmed SARS-CoV-2 infection as determined by FDA-approved rapid diagnostic (e.g., polymerase chain reaction [PCR]) assay within the preceding 7 days (168 hours).
* Has at least 2 COVID-19 related symptoms on the 14-question COVID-19 questionnaire.
* Has peripheral capillary oxygen saturation (SpO2) >93% by pulse oximetry.
* C-reactive protein (CRP) >50 mg/L or lymphopenia (<1.5×109/L) or neutrophilia (>7.5×109/L).
* Agrees to the collection of blood and urine samples, nasal swabs , and non-invasive oxygen monitoring (via pulse oximeter) per protocol.
* Willing to receive 4 injections at separate sites on the thigh or abdomen.
* Women of childbearing potential must agree to either abstinence or use of at least one primary form of contraception (not including hormonal contraception) from the time of screening through Day 29 following randomization.
* Agrees to not participate in any other clinical trial (both pharmacologic and other types of interventions) through Day 29 following randomization

Exclusion Criteria:

* Received or contemplating any COVID-19 vaccine or participated in a COVID-19 vaccine trial.
* Subject is considered to be in their last few weeks of life prior to this acute illness.
* History of pulmonary alveolar proteinosis.
* History of hematopoietic stem cell transplant or solid organ transplant.
* Previous malignancy and lymphoproliferative disorders (within the last 5 years) with the exception of stable prostate cancer and basal cell carcinoma.
* Chronic obstructive pulmonary disease on long-term oxygen therapy - subjects with forced expiratory volume in 1 second known to be <50% will also be excluded.
* Demyelinating disease.
* Known history of hepatitis B, HIV, or untreated hepatitis C infection
* Severe hepatic impairment or known cirrhosis - Child-Pugh score B or higher.
* Acute kidney injury Stage 3
* Tuberculosis or other severe infections such as (non-COVID-19) sepsis, abscesses, fungal superinfection and opportunistic infections requiring treatment.
* Positive Quantiferon Gold test at screening
* Moderate or severe heart failure (New York Heart Association Class III/IV).
* Treatment with monoclonal antibodies targeting cytokines (e.g., TNF inhibitors [adalimumab, infliximab, etanercept, golimumab, certolizumab]; anti-IL-1 [e.g., anakinra, canakinumab]; anti-IL-6 or anti-IL-6r [e.g., tocilizumab, sarilumab, sitlukimab]; or T-cells [e.g., abatacept]) in past 90 days (5 half-lives of the drug), or contemplating treatment with any of these agents during the trial period.
* Treatment with monoclonal antibodies targeting B-cells (e.g., rituximab, and including any targeting multiple cell lines including B-cells) in the 3 months prior to screening.
* Received GM-CSF agents (e.g., sargramostim) within 2 months prior to screening.
* Treatment with other immunosuppressants in the 4 weeks prior to screening and in the judgment of the Investigator, the risk of immunosuppression with adalimumab is larger than the risk of COVID-19.
* Treatment with small molecule tyrosine kinase inhibitors (e.g., baricitinib, ibrutinib, acalabrutinib, imatinib, gefitinib), in the 4 weeks prior to screening.
* Received or contemplating receipt of any live vaccine or any investigational vaccine in the 4 weeks prior to screening.
* Current participation or previous participation in any other clinical trial within 30 days prior to randomization.
* Subjects with known hypersensitivity to adalimumab or excipients of adalimumab as stated in the label.
* Pregnant female
* Lactating female
* Women of childbearing potential who do not agree to either abstinence or use of at least one primary form of contraception (not including hormonal contraception) from the time of screening through Day 29 following randomization.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Establish whether treatment with adalimumab is associated with a lower rate of progression to severe disease as defined by severe illness or critical illness, or death in outpatient subjects with COVID-19 | 28 Days
  Proportion of subjects with the following outcomes attributed to COVID-19 from time of first dose through Day 28 following randomization:
  * Death
  * Alive and hospitalized or requiring supplemental oxygen for ≥1 hour
  * Alive and not hospitalized or requiring supplemental oxygen for ≥1 hour
Assess the safety of adalimumab in subjects with COVID-19 | 28 Days
  Incidence of Grade 3 and Grade 4 clinical adverse events (AEs) from first dose through Day 28 following randomization

SECONDARY OUTCOMES:
Assess the impact of treatment with adalimumab on clinical course of COVID-19 infection | 120 Days
  Clinical status by 9-point WHO COVID 19 ordinal scale from first dose through Day 120 following randomization
  * Incidence of venous thromboembolism, CVA, myocardial infarction, and acute kidney injury C from first dose through Day 120 following randomization
  * Time to resolution of symptoms using 14 point COVID-19 Symptom Score from first dose through Day 120 following randomization
  * COVID-19 Clinical Assessment from first dose through Day 120 following randomization

IPD SHARING:
Plan to Share IPD: No